CLINICAL TRIAL: NCT03943030
Title: Effects of Pulmonary Rehabilitation on Cardiovascular Parameters in Patients With COPD
Brief Title: Cardiovascular Effects of Pulmonary Rehabilitation in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 96766418100005327
Record Dates: First submitted 2019-01-26; First posted 2019-05-09 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Pulmonary rehabilitation; Chronic Obstructive Pulmonary Disease; Cardiovascular effects; Endothelial dysfunction
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial, performed with two groups: intervention and controls (usual care).
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulmonary rehabilitation (Experimental): The PR program will consist of supervised physical exercise sessions, which will be held 3 times a week for 8 weeks, and weekly educational sessions. Exercise sessions include aerobic exercise (30 min to 45 min) and lower limb and upper limb strength training, as well as warm-up and muscle stretching exercises after exercise. The exercise load will be individualized and determined from the patients' baseline tests, being increased progressively throughout the sessions. A baseline evaluation will be performed, which will be repeated after 9 weeks, including: clinical and laboratory parameters, endothelial function (FMD) and brachial ankle index (ABI) and exercise tests. Outcomes usually used in the assistance to evaluate PR will also be measured.
  Interventions: Other: Pulmonary rehabilitation
- Group control (No Intervention): The group will not receive pulmonary rehabilitation intervention. Patients will be guided and maintain their daily and routine lives normally during the evaluation process. However, a baseline evaluation will be performed, which will be repeated after 9 weeks: clinical and laboratory parameters, endothelial function (FMD) and brachial ankle index (ABI) and exercise tests. Outcomes commonly used in the assistance to assess PR will also be measured.

INTERVENTIONS:
Other: Pulmonary rehabilitation — The PR program will consist of supervised physical exercise sessions, which will be held 3 times a week for 8 weeks, and weekly educational sessions. Exercise sessions include aerobic exercise (30 min to 45 min) and lower limb and upper limb strength training, as well as warm-up and muscle stretching exercises after exercise. The exercise load will be individualized and determined from the patients' baseline tests, being increased progressively throughout the sessions. A baseline evaluation will be performed, which will be repeated after 9 weeks, including: clinical and laboratory parameters, endothelial function (FMD) and brachial ankle index (ABI) and exercise tests. Outcomes usually used in the assistance to evaluate PR will also be measured.
  Arms: Pulmonary rehabilitation

SUMMARY:
Introduction: Chronic obstructive pulmonary disease (COPD) is characterized by airflow obstruction, which is clinically manifested by dyspnea and leads the patient to a vicious cycle of sedentary lifestyle. Pulmonary rehabilitation (PR) is an important therapeutic strategy to break this cycle. Cardiovascular diseases are frequent in patients with (COPD) and are associated with higher mortality. The effects of (PR) on cardiovascular risk factors in patients with (COPD) have been little studied so far. Objectives: To evaluate the effects of pulmonary rehabilitation compared to the control group on cardiovascular risk factors in patients with (COPD). Methods: A randomized clinical trial will be conducted. Patients with (COPD) will be divided into two groups: Group I (GI): group that will be rehabilitated, with 3 weekly sessions, for 8 weeks and Group II (GII): control group, without intervention. In both groups, a baseline evaluation will be performed, which will be repeated after 9 weeks and consists of: clinical and laboratory parameters, endothelial function (FMD) and brachial ankle index (ABI). Outcomes commonly used in the assistance to assess (PR) will also be measured. Expected Results: The study is expected to improve understanding of the impact of (PR) on cardiovascular variables in patients with (COPD).

DETAILED DESCRIPTION:
Measures and instruments Before the rehabilitation program, a baseline evaluation will be performed, which will include: anthropometric evaluation, Framingham cardiovascular risk score calculation, (mMRC) scale completion, and International Physical Activity Questionnaire (IPAQ). Baseline lung function data will be obtained from patients' medical records. The severity of (COPD) will be determined by spirometric classification of the Gold consensus, Body-mass index, airflow obstruction, dyspnea, and exercise (BODE) and Gold (ABCD) scale. To evaluate exercise capacity, a 6-minute (s) walk test (6MWT), an incremental cardiopulmonary exercise test (ECT) on a cycle ergometer, and a cardiopulmonary exercise test with a constant load on a cycle ergometer will be performed. All patients will undergo evaluation of endothelial function and (ABI) (brachial ankle index). Laboratory tests, exercise tests, evaluation of endothelial function and (ABI) will be performed before and after the pulmonary rehabilitation program. Two visits will be necessary to carry out the tests: on the first visit blood will be collected for laboratory tests, the questionnaires will be answered, anthropometric data collected and the incremental (ECP) will be performed; at the second visit, the (ABI) and endothelial function will be measured and the constant load (TECP) will be performed. There will be a minimum of 48 hours between visits. The incremental (ECP) will be performed only at baseline. In the anthropometric evaluation will be determined the weight and the height, being calculated the body mass index through the formula; weight (kg) / height2 (m). Laboratory Tests Total cholesterol and fractions, triglycerides, C-reactive protein, fasting glycemia, Glutamic oxaloacetic transaminase (GOT), Glutamic-pyruvic transaminase (GPT), urea and creatinine and protein C will be collected baseline and after intervention. Pulmonary function Results of spirometry, pulmonary diffusion by carbon monoxide (DLco) and lung volumes (plethysmography) will be recorded, which are performed in the care routine and will be obtained from the patients' records. Exercise tests The (6MWT) will be performed in a 30 meter corridor, with continuous monitoring of peripheral oxygen saturation (SpO2) and heart rate. Before and after the test the respiratory rate and the intensity of the dyspnea will be determined. The distance covered in 6 minutes will be recorded. The test will be performed in accordance with the guidelines and predicted values previously described. The maximum incremental (TECP) limited by symptoms will be performed on an electromagnetic bicycle using a ramp protocol. After 2 minutes of standing monitoring, the patient will pedal for 2 minutes without load. The load ramp will be individualized so that the incremental test lasts between 8 and 12 minutes. The incremental (TECP) will be performed according to the recommendations of the. The constant load test will be performed with 75% of the maximum load reached in the incremental (TECP). During the tests performed on the exercise bicycle, the electrocardiographic tracing and (SpO2) will be continuously monitored. Significant desaturation will be considered when (SpO2) falls ≥ 3%. Endothelial function will be non-invasively assessed by flow-mediated dilatation in the brachial artery using a high-resolution ultrasound imaging device (SONOSITE®, M-Turbo, Sony). Brachial ankle index, the assessment of the systolic arterial pressure of the brachial arteries and posterior tibial arteries will be performed bilaterally using a portable vascular Doppler, with a sphygmomanometer positioned 3 cm above the cubital fossa in the upper limbs and 3 cm above the medial malleolus in the lower limbs. The randomization will be performed through an online software at www.random.org, then will be stored in a stealth location. A blinded investigator will generate a numerical sequence of the randomized patients who meet the eligibility criteria. The study was not done with the total number of patients diagnosed with (COPD). Those divided into two groups: intervention and control.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of COPD, in stages II, III and IV, according to criteria of the Global Initiative for COPD;
* Stable patients (no exacerbation in the last 4 weeks).

Exclusion Criteria:

* Patients with contraindications to exercise (decompensated ischemic heart disease or neuromuscular diseases) or unable to perform evaluations and / or participate in the pulmonary rehabilitation program.
* Bood pressure greater than 160/90 mmHg,
* Serum cholesterol greater than 220,
* Diabetes mellitus,
* Active smoking or using vasodilator drugs (calcium channel blockers and ACE inhibitors).
* Use of β-blocker will be directed to ingest the last dose of this drug 24 hours before the measurement of endothelial function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2021-12-18 (Actual); Study Completion 2023-07-18 (Actual)

PRIMARY OUTCOMES:
Dilatation mediated by the flow of the brachial artery | Eight Weeks.
  The flow-mediated dilatation of the brachial artery will be assessed non-invasively by the ultrasound device (SONOSITE®, M-Turbo, Sony). A high-frequency transducer (HFL38xp, SONOSITE®, Sony) will be used to obtain longitudinal images of the brachial artery walls.

SECONDARY OUTCOMES:
Brachial ankle index | Eight Weeks.
  The calibration of the brachial, pediatric and posterior tibial arteries bilaterally will be performed using a portable vascular Doppler.
Body-mass Index | Eight Weeks.
  Evaluate the weight of a person in relation to their height.
Airflow Obstruction | Eight Weeks.
  Pulmonary function through spirometry, that allows to measure forced expiratory volume in the first second. It's the maximum expired volume at the first second of an maximum expiration.
Dyspnea - Modified Medical Research Council (mMRC scale) | Eight Weeks.
  Evaluates dyspnea intensity, ranging from zero to four:
  Grade 0 - No troubled by breathlessness except on strenous exercise. Grade 1 - Short of breath when hurryng or walking up a slight hill. Grade 2 - Walks slower than contemporaries on the level because of breathlessness or has to stop for breath when walking at own pace.
  Grade 3 - Stops of breath after walking 100m or after a few minutes on the level.
  Grade 4 - Too breathless to leave the house or breathless when dressing or undressing.
  The scale is gradual according to the patient's dyspnea level
Exercise Capacity | Eight Weeks.
  Distance traveled on the 6-min walk tes (6MWT).
Laboratory Tests - Total cholesterol | Eight Weeks.
  Blood collection to measure total cholesterol performed at HCPA.
Laboratory Tests - HDL cholesterol | Eight Weeks.
  Blood collection to measure HDL cholesterol performed at HCPA.
Laboratory Tests - LDL cholesterol | Eight Weeks.
  Blood collection to measure LDL cholesterol performed at HCPA.
Laboratory Tests - Triglycerides | Eight Weeks.
  Blood collection to measure triglycerides performed at HCPA.
Laboratory Tests - C-reactive protein | Eight Weeks.
  Blood collection to measure C-reactive protein performed at HCPA.
Laboratory Tests - Glutamic oxaloacetic transaminase (GOT) | Eight Weeks.
  Blood collection to measure GOT performed at HCPA.
Laboratory Tests - Glutamic-pyruvic transaminase (GPT) | Eight Weeks.
  Blood collection to measure GPT performed at HCPA.
Laboratory Tests - Urea | Eight Weeks.
  Blood collection to measure Urea performed at HCPA.
Laboratory Tests - Creatinine | Eight Weeks.
  Blood collection to measure creatinine performed at HCPA.
Anthropometric evaluation - Waist circumference | Eight Weeks.
  The position the tape measure at the point between the last rib and the iliac crest with the smallest measure.
Anthropometric evaluation - Circumference of the hip | Eight Weeks.
  Twill be measured with a tape measure at the highest measurement on the hip.

CONTACTS AND LOCATIONS:
Overall Officials: Marli Knorst, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No